CLINICAL TRIAL: NCT03296761
Title: Endothelial Cell Specific Molecule-1 (ESM-1): a Novel Biomarker for ARDS Endothelial Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jingyuan,Xu (Other)
Responsible Party: Sponsor-Investigator, Jingyuan,Xu, chief doctor, Southeast University, China
Organization: Southeast University, China (Other)
Other Study IDs: 2017ZDSYLL081-P01
Record Dates: First submitted 2017-09-25; First posted 2017-09-28 (Actual); Last update posted 2017-11-01 (Actual); Status verified 2017-09

CONDITIONS: Evaluate the Correlation Between the Level of ESM-1 and the Prognosis of the Patients With ARDS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ESM-1<5ng/ml
- ESM-1≥5ng/ml

SUMMARY:
To observe the changes of plasma ESM-1 levels in patients with ARDS, and to explore its clinical significance.

DETAILED DESCRIPTION:
70 patients who diagnosed as ARDS were included in this study. Then keep blood samples from these patients in the first day, the third day and the seventh day, detect ESM-1 level in plasma by ELISA. Record Severity of illness and survival status of every patient within 28 days. Objective to evaluate the correlation between the level of ESM-1 in plasma and the prognosis of the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted to ICU diagnosed of ARDS (Berlin definition）in 48h
2. Patients age between 18 years old and 80 years.

Exclusion Criteria：

1. Pregnant women,
2. Patients with malignant tumor,
3. Immunosuppression or immunocompromised patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population admitted to ICU of Zhongda hospital ，diagnosed of ARDS
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2017-12-20 (Estimated); Study Completion 2018-02-20 (Estimated)

PRIMARY OUTCOMES:
mortality | 28-day

CONTACTS AND LOCATIONS:
Overall Officials: Haibo qiu, Study Chair — Zhong-Da Hospital, School of Medicine, Southeast University,
Locations (1):
- Nanjing Zhongda Hospital, School of Medicine, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No